CLINICAL TRIAL: NCT06847126
Title: Comparison of Empirical Intravenous Beta-Lactam Antimicrobials Plus Metronidazole and Oral Cefixime Plus Metronidazole Therapy for the Treatment of Liver Abscess: an Open Label Randomized Controlled Clinical Trial
Brief Title: Empirical Intravenous Beta-Lactam Plus Metronidazole Vs Oral Cefixime Plus Metronidazole for the Treatment of Liver Abscess
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Deba Prasad Dhibar, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEC-INT/2025/Study-2667
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Liver Abscess
Keywords: Liver Abscess, Empirical antimicrobials, Beta-lactam antimicrobials, Intravenous, Oral, Cefixime, Metronidazole
MeSH Terms: conditions — Liver Abscess | interventions — WW Domain-Containing Oxidoreductase; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Beta-Lactam antimicrobials (Active Comparator): Intravenous beta-lactam antimicrobial for 2 weeks Plus Intravenous Metronidazole (750 mg q 8 hourly) for 2 weeks and standard care
  Interventions: Drug: Intravenous beta-lactam antimicrobial for 2 weeks Plus Intravenous Metronidazole (750 mg q 8 hourly) for 2 weeks; Other: Standard medical care
- Oral Cefixime (Active Comparator): Tablet Cefixime (200 mg q 12 hourly) for 2 weeks Plus Table Metronidazole (800 mg q 8 hourly) for 2 weeks and standard care
  Interventions: Drug: Tablet Cefixime (200 mg q 12 hourly) for 2 weeks Plus Tablet Metronidazole (800 mg q 8 hourly) for 2 weeks; Other: Standard medical care

INTERVENTIONS:
Drug: Intravenous beta-lactam antimicrobial for 2 weeks Plus Intravenous Metronidazole (750 mg q 8 hourly) for 2 weeks — Intravenous beta-lactam antimicrobial for 2 weeks Plus Intravenous Metronidazole (750 mg q 8 hourly) for 2 weeks and standard care
  Other Names: Standard care
  Arms: Intravenous Beta-Lactam antimicrobials
Drug: Tablet Cefixime (200 mg q 12 hourly) for 2 weeks Plus Tablet Metronidazole (800 mg q 8 hourly) for 2 weeks — Tablet Cefixime (200 mg q 12 hourly) for 2 weeks Plus Tablet Metronidazole (800 mg q 8 hourly) for 2 weeks
  Other Names: Standard Medical care
  Arms: Oral Cefixime
Other: Standard medical care — Percutaneous drainage or aspiration of the abscess along resuscitative and symptomatic medications

SUMMARY:
Liver abscess (LA) is potentially life threatening medical emergency requiring prompt medical intervention. The backbone of therapy is prompt empirical antimicrobial with or without percutaneous drainage/ aspiration of the abscess. The standard care for liver abscess includes empirical antimicrobials consisting both antibacterial and amoebicidal agents along with percutaneous drainage or aspiration of the collection. The antimicrobial regimen should cover against E. histolytica until microbial etiology is established or liver abscess of amoebic etiology is ruled out. But still there is no straightforward general agreement or evidence based on clinical studies regarding the standard protocol for empirical antimicrobials concerning choice, route of administration or duration of antimicrobials therapy. Most of the experts preferred intravenous antimicrobials over oral antimicrobials for the treatment of liver abscess with or without complication. But, there is no clinical trial evidence to support the rational of using intravenous antibiotics up front instead of oral antimicrobials. Recently published institutional study also suggested that empirical oral antimicrobials (Cefexime/Ciprofloxacin) were efficacious for the treatment of uncomplicated liver abscess, successfully managing around 90 % cases of liver abscess. When treating a liver abscess, the choice of antimicrobials and the administration technique must be specially tailored depending upon the existence of complications and the patient's clinical reaction. In the absence of clinical trials, the rational for using of intravenous broad spectrum antibiotics upfront instead of oral antimicrobials for the treatment of liver abscess with or without complications is doubtful and may appear injudicious contributing future rise of antimicrobial resistance. The use of intravenous antibiotics upfront may also unnecessarily lengthen hospital stays, enhance therapeutic expenditure, and raise the risk of hospital-acquired infections in patients who are capable for taking antimicrobials orally. Oral antimicrobials strategy will promote earlier discharge from the hospital and the patient can return to usual activities earlier. This study aims to provide valuable insights into the comparison and efficacy of empirical intravenous Beta-lactam antimicrobials plus Metronidazole and oral Cefixime plus Metronidazole therapy for the treatment of uncomplicated liver abscess. In this randomised controlled open label clinical trial all the patients with newly diagnosed liver abscess confirmed with radiology imaging, either by USG or CT scan, presenting at emergency or medical OPD will be screened for enrolment in the study. Following written informed consent from the participants and/or their legal guardian, those who meet the inclusion and exclusion criteria will be recruited in the study. Subsequently the participants will be randomized into either intravenous or oral antimicrobial group. The intravenous-group will receive Beta-lactam antimicrobials (i.e Piperacillin-Tazobactum 4.5g q 8 hourly or Ceftriaxone 1g q 12 hourly or Meropenem 1g q 8 hourly or Imipenem-Cilastatin 500mg q 6 hourly) Plus intravenous Metronidazole 750mg q 8 hourly for 2weeks. The oral-group will receive tablet Cefixime 200 mg q 12 hourly plus tablet Metronidazole 800 mg q 8 hourly for 2 weeks. Both the group will be provided standard care of therapy including percutaneous drainage or aspiration as per indication and will be followed up for 8 weeks. The primary outcome of clinical cure and secondary outcome of incidence of treatment failure, mortality, duration of antimicrobial therapy, recurrence, adverse drug reaction (ADR), complications will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria: All symptomatic patients with liver abscess verified by radiological imaging, either by computed tomography (CT) scan or ultrasound (USG), regardless of gender (male or female) and age ≥ 18 years, will be screened for registration in the study.

-

Exclusion Criteria: Patients with past history of liver abscess, chronic kidney disease (CKD), hypersensitivity to either Metronidazole or Cefixime or Beta-lactam antimicrobials will not be allowed to participate in the study. Patients with organ dysfunction with shock (blood pressure < 90/60 mmHg), acute respiratory distress syndrome requiring oxygen therapy (PaO2/FiO2 ≤ 300 or SpO2 ≤92%), encephalopathy (altered sensorium with GCS < 15), acute kidney injury (increase in serum creatinine to ≥ 1.5 times from the baseline or serum creatinine ≥ 1.5) and not able to take orally will not be considered for participation in the study. Patients who are pregnant, have already received antimicrobials for more than 48 hours before to admission, or are receiving blood thinners such as antiplatelets or anticoagulants within 4 weeks of presentation and are unwilling to provide informed consent will also be excluded from the trial.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | 8 weeks
  "clinical cure" is defined as defined as participants becoming asymptomatic with fever resolution for ≥48 hours, including USG demonstrating no drainable or aspiratable collection in the liver along with removal of the pigtail catheter if any.
Treatment failure | 8 weeks
  "Treatment failure" is defined as the fulfilling of any one or more of the following conditions:
  1. Persistently symptomatic even after 72 h of empirical antimicrobial therapy and percutaneous aspiration or drainage of the hepatic collection
  2. Emergence of fresh or additional collection in the liver during the course of empirical antimicrobial therapy
  3. Emergence of shock and or new onset organ failure (Encephalopathy, ARDS, AKI, MODS) during the course of therapy, leading to modification of oral antimicrobials to intravenous antimicrobials or up gradation of the ongoing intravenous antimicrobials
  4. If pus culture demonstrates growth of microorganism which is not sensitive to the ongoing antimicrobials (intravenous Beta-lactam or oral Cefixime) along with inadequate clinical response to the therapy
  5. Participants requiring persistent drainage or repeated aspiration of the abscess even after 4 weeks of empirical antimicrobial therapy

SECONDARY OUTCOMES:
Duration of the therapy | 8 weeks
  Number of days of empirical antimicrobial therapy is required to achieve clinical cure
Need for prolong antibiotics therapy | 8 weeks
  Asymptomatic participants requiring persistent drainage or repeated aspiration of the abscess even after 2 weeks of empirical antimicrobial therapy to achieve clinical cure
Duration of hospital stay | 8 weeks
  Number of days receiving in-hospital medical care
Readmission | 8 weeks
  Participants requiring repeated admission with in-hospital medical care to achieve clinical
Recurrence of liver abscess | 8 weeks
  Emergence of new liver abscess after achieving clinical cure during 8 weeks of follow up
Adverse drug reaction (ADR) | 8 weeks
  Incidence of adverse drug reaction related to the ongoing antimicrobial therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research (PGIMER), Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
Plans to share individual participant data (IPD) will considered with reasonable request to the principal investigator depending upon Institutional Ethic Committee approval.